CLINICAL TRIAL: NCT04324502
Title: Mobile Application to Collect PRO Data in NET Patients
Status: Recruiting | Type: Observational
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: Ampersand Health Ltd (Unknown); Neuroendocrine Cancer UK (Unknown)
Responsible Party: Sponsor
Other Study IDs: 259461
Record Dates: First submitted 2020-03-25; First posted 2020-03-27 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-03

CONDITIONS: Neuroendocrine Neoplasms (Tumours)
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neuroendocrine neoplasms (tumours): Patients with a diagnosis of neuroendocrine neoplasm who are due to undergo one of the following treatments: chemotherapy, everolimus, sunitinib, somatostatin analogues, peptide receptor targeted therapy, embolization/ ablative therapies or surgery.

SUMMARY:
Observational trial to assess the feasibility of monitoring patient reporting symptoms via mobile devices

DETAILED DESCRIPTION:
Neuroendocrine tumours (NET) are uncommon cancers with varied presentation. Patients are treated in specialist centres, and may sometimes have up to 4 lines of treatment; with the attendant complications. To date there has been no study capturing precisely patient reported outcomes (PROMs) and changes in QoL post treatment.

We have worked with the national patient charity and support group (Neuroendocrine Tumour Patient Foundation) and UKINETS, to develop a mobile application that will allow patients to capture details of their symptoms, as well as changes to quality of life during and post treatment. The application has been designed as an aide to patients, capturing details of their illness, treatment and interaction with the healthcare team (appointments).

This study aims to assess whether use of mobile app technology is helpful for patients undergoing medical and surgical therapy for neuroendocrine tumours. The trial is non-invasive and allows participants to record daily symptoms and raise alerts whilst they are undergoing different therapies. Health related quality of life during therapy will be assessed at specified times using EORTC validated questionnaires. The study also aims to investigate any difference in clinicians' response to PROMs; and the time taken to institute change, in any.

Participants are able to download the application from their mobile device app store from whichever location they wish, provided that they have regular internet access to download the app. Participants will be asked to provide daily responses pertaining to their health outcomes (PROs) in addition to completing validated quality of life questionnaires (EORTC CLQ - C30 and EORTC GINET21) at regular intervals over a 4 year period, prior to their treatment starting and throughout their treatment (months 0,3,6,12; and 6 monthly thereafter). This data will be stored in a research-specific database of de-identified patient-reported outcomes on quality of life and health.There are added features for participants to enter their medication information and appointments in the outpatient clinic; functionality to set reminders to take their medication; as well as reminders for upcoming hospital visits; and links to email addresses to contact their primary care teams. Clinicians are able to access the data to identify problems and track response to interventions.

The data will be stored in an encrypted format on the secure servers of Ampersand Health Ltd, who will export the data to the Chief Investigator at King's College Hospital at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of a NET
* Planned treatment for NET
* Able to give informed consent
* Able to understand the language of the questionnaires
* A minimum expected survival of 6 months
* All performance status is acceptable
* 18 years of age or over

Exclusion Criteria:

* Concurrent malignancies for which they are undergoing treatment
* No smartphone / device
* Any physical, psychological or comprehension problems that prevents completion of questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of neuroendocrine neoplasm who are due to undergo one of the following treatments: chemotherapy, everolimus, sunitinib, somatostatin analogues, peptide receptor targeted therapy, embolization/ ablative therapies or surgery.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-07-20 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Reporting compliance | 4 years
  The primary endpoint is patient reporting compliance, defined as the number of days with any patient report submitted during the course of treatment. This will be unique to each course of therapy since they have different durations of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- King's College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF